CLINICAL TRIAL: NCT05398913
Title: Effects of Rimonabant on Walking Abilities in Incomplete Spinal Cord Injury: a Proof-of-concept Study
Brief Title: Effects of Rimonabant on Walking Abilities in Incomplete Spinal Cord Injury
Acronym: RIMOFATSCI-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Principal Investigator, Antonio Oliviero, Principal Investigator, Hospital Nacional de Parapléjicos de Toledo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FHNP-CT002
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal cord injury; Walking endurance; Incomplete SCI; Traumatic
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rimonabant

STUDY DESIGN:
Intervention Model Description: Randomized crossover study with three arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Two pills of placebo will be administered for 5 consecutive days, once per day.
  Interventions: Drug: Rimonabant
- Rimonabant 2.5 mg (Active Comparator): One pill of placebo and one pill of Rimonabant 2.5mg will be administered for 5 consecutive days, once per day.
  Interventions: Drug: Rimonabant
- Rimonabant 5 mg (Active Comparator): Two pills of Rimonabant 2.5mg will be administered for 5 consecutive days, once per day.
  Interventions: Drug: Rimonabant

INTERVENTIONS:
Drug: Rimonabant — Rimonabant

SUMMARY:
Randomized placebo-controlled safety and feasibility study with crossover design (3 arms). Placebo or Rimonabant 2.5mg or Rimonabant 5mg will be administered for 5 days. Exploratory efficacy will be tested using six-min walking test.

DETAILED DESCRIPTION:
Randomized placebo-controlled safety and feasibility study with crossover design (3 arms). Placebo or Rimonabant 2.5mg or Rimonabant 5mg will be administered for 5 days. Exploratory efficacy will be tested using six-min walking test.

Main goal is to test safety of Rimonabant in a specific population (incomplete spinal cord injury).

ELIGIBILITY:
Inclusion Criteria:

* Traumatic spinal cord injury
* Incomplete lesion (AIS D)
* Neurological level between C4 and L1
* Chronic stage (>1 year since injury)
* Preserved walking ability for at least 5 m (aid allowed)
* Psychiatric assessment to exclude individuals with high suicide risk
* Capability to provide informed consent
* For fertile women, possibility to use anti conceptive methods

Exclusion Criteria:

* Non traumatic spinal cord injury
* AIS A, B, C or E
* Neurological level above C4 or below L1
* Subacute stage (<1 year since injury)
* Preserved walking ability for less than 5 m (aid allowed)
* Pregnancy or breast feeding
* For fertile women, impossibility to use anti conceptive methods
* Anticoagulant treatment
* Hypothyroidism
* Severe kidney or liver dysfunction
* Severe depression
* Fatigue treatment in the last 6 months
* Impossibility to reach the Hospital
* Impossibility to provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Adverse events (safety) | 150 days
  number of AE
6 min walking test (efficacy) | 5 days
  6 min walking test (meters and number of stops are reported)
Biochemical and urine analysis (safety) | 8 days
  Number of participants with clinically significant abnormal laboratory tests results
ECG (safety) | 8 days
  Number of participants with clinically significant abnormal ECG readings
Beck Depression Inventory (BDI) (safety) | 15 days
  Range 0-63 (higher values more severe)
Hospital Anxiety and Depression Scale (HAD) (safety) | 15 days
  Range 0-21(higher values more severe)
Modified Ashworth Scale (safety) | 15 days
  Range 0-4 (higher values more severe)
Penn Scale (safety) | 15 days
  Range 0-4 (higher values more severe)

SECONDARY OUTCOMES:
10 m test (efficacy) | 5 days and 15 days
  Time to walk 10 m (no stops are allowed)
6 min walking test (efficacy) | 15 days
  6 min walking test (meters and number of stops are reported)
Borg Scale (efficacy) | 5 days and 15 days
  Borg Scale punctuation after 6 min waking test. Range 0-10.
WISCI II (efficacy) | 5 and 15 days
  Range 0-20 (higher values less severe)
Motor Score (efficacy) | 8 days
  Motor Score (ISNCSCI). Range 0-20 (higher values less severe)
Fatigue Severity Scale (FSS) (Efficacy) | 5 and 15 days
  FSS puntuación. Range 0-7 (higher values more severe)
European Quality of Life -5 Dimensions (EQ-5D) (efficacy) | 8 days
  EQ-5D questionnaires have 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 3 problem levels corresponding to patient response choices (higher values worst). A quality-of-life score is obtained according to the answers to the questionnaires (algorithm to calculate the score in euroqol.org). The maximum score is 1 that indicates excellent quality of life (range for Spanish version 0.5-1).
Patient global impression of changes (PGIC) (efficacy) | 5 and 15 days
  PGIG score. Range 1-7 (higher values indicate worsening)
Pain numeric rating scale | 8 days
  Range 0-10 (higher values more severe)
Health state visual analogically scale | 8 days
  Range 0-100 mm (higher values indicate higher health state )

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Oliviero, MD, PhD, Principal Investigator — Hospital Nacional de Parapléjicos
Locations (1):
- Hospital Nacional de Paraplejicos, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request